CLINICAL TRIAL: NCT04056806
Title: A Prospective, Randomized Controlled Trial of 2- Day vs. 5- Day Terlipressin and Ceftriaxone in the Prevention of Very Early Rebleeding in Patients With Acute Gastroesophageal Variceal Hemorrhage
Brief Title: 2- Day vs. 5- Day Terlipressin and Ceftriaxone in the Control Acute Gastroesophageal Variceal Hemorrhage
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: E-DA Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMRP39107N
Record Dates: First submitted 2019-08-06; First posted 2019-08-14 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Variceal Rebleeding Rate and Infections
MeSH Terms: conditions — Infections | interventions — Terlipressin; Powders

STUDY DESIGN:
Intervention Model Description: A prospective, randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): receiving terlipressin 2mg bolus on enrollment followed by 1mg per 6 hours. Both Terlipressin infusion and Ceftriaxone continue till 48 hours after endoscopic therapy
  Interventions: Drug: Terlipressin 1Mg Powder for Conventional Release Solution for Injection Vial
- Gruoup B (Active Comparator): receiving terlipressin 2mg bolus instituted on enrollment followed by 1mg per 6 hours. Ceftriaxone 1gm intravenously dose of ceftriaxone 1gm at 24 h interval. Both Terlipressin infusion and Ceftriaxone continue till 5 days after endoscopic therapy.
  Interventions: Drug: Terlipressin 1Mg Powder for Conventional Release Solution for Injection Vial

INTERVENTIONS:
Drug: Terlipressin 1Mg Powder for Conventional Release Solution for Injection Vial — efficacy comparison between 2 days and 5 days
  Other Names: Ceftriaxone 1gm

SUMMARY:
The use of prophylactic antibiotics in cirrhotics with gastrointestinal bleeding has been a routine clinical practice . It is still unknown whether use of short term vasoconstrictors and antibiotics could have superior acute hemostatic rate.

Thus, the investigators conducted a trial to compare the effectiveness between participants receiving terlipressin and ceftriaxone 5 days and terlipressin and ceftriaxone 2 days after endoscopic therapy in cirrhotic patients presenting with acute gastro-esophageal variceal hemorrhage..

DETAILED DESCRIPTION:
Acute gastro-esophageal variceal hemorrhage is a dreadful complication of portal hypertension. Meta-analysis showed that the combination of vasoconstrictor and endoscopic therapy is superior to endoscopic therapy or vasoconstrictor alone in the control of acute esophageal variceal hemorrhage. Bacterial infections are frequently encountered in cirrhotic patients presenting with acute upper gastrointestinal bleeding. The association of bacterial infections to variceal bleeding may increase the occurrence of variceal rebleeding and mortality. A study has shown that antibiotic prophylaxis in patients with acute esophageal variceal hemorrhage may reduce infection as well as prevent rebleeding. Currently, most guidelines recommend that vasoactive drugs should be continued for 3 to 5 days after endoscopic therapy and antibiotics should be instituted for up to 7 days to manage patients with acute esophageal variceal hemorrhage . On the other hand, some studies in recent years implied that short term vasoconstrictors or antibiotics could achieve similar low variceal rebleeding rates. The use of prophylactic antibiotics in cirrhotics with gastrointestinal bleeding for only one single dose or 3 days appeared to be feasible. It is still unknown whether use of short term both vasoconstrictors and antibiotics could have similar acute hemostatic rate.

Thus, the investigators conducted a trial to compare the effectiveness between participants receiving terlipressin and ceftriaxone 5 days and terlipressin and ceftriaxone 2 days after endoscopic therapy in cirrhotic patients presenting with acute gastroesophageal variceal hemorrhage..

ELIGIBILITY:
Inclusion Criteria:

1. Patients were diagnosed to have cirrhosis based on history, physical examinations, image studies or histological examination..
2. Age ranges between 20-80 y/o.
3. Patients presenting with hematemesis and /or melena within 24 hours of inclusion.
4. Esophageal variceal bleeding is controlled by esophageal variceal ligation (EVL). Gastric variceal bleeding is controlled by endoscopic glue ( histoacryl) injection.

   -

Exclusion Criteria:

1. Uncertain of bleeding source.
2. Failure in endoscopic therapy.
3. Had variceal bleeding or peptic ulcer bleeding in recent one month
4. has evidence of bacterial infections or possible infection at entry ( such as fever > 37.5。 C, white blood cells> 10000/cumm, urine leukocytes >10/ field, pneumonic patches on chest x-ray, ascitic polymorphonuclear cells > 250/cumm, cellulitis or other focal infections).

2) ever received antibiotics within 4 weeks before index upper gastrointestinal bleeding.

3) presence of cardiopulmonary embarrassment 4) association with uremia and receiving hemodialysis or peritoneal dialysis. 5) presence of deep jaundice (serum bilirubin > 10 mg/dl), hepatic encephalopathy stage III or IV, massive or refractory ascites 6) presence of chronic kidney disease ( serum creatinine > 2 mg/dl) or hepatorenal syndrome 7) Had history of cerebrovascular accident, coronary artery disease, complete AV block or peripheral vascular disorder 6) association with human immunodeficiency virus (HIV) infection, advanced carcinoma or hepatocellular carcinoma Barcelona Club Liver Cancer (BCLC) class C or D.

7) allergy to terlipressin, cephalosporins or penicillin 8) pregnancy. 9) Uncooperative or decline to be enrolled

-

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-08 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
incidence of very early rebleeding | 5 days
  The occurrence of variceal rebleeding after initial hemostasis

SECONDARY OUTCOMES:
Bacterial infections, 42-day rebleeding, mortality | 6 weeks
  Incidence of bacterial infections & rebleeding, mortality in 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- E-Da Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No